CLINICAL TRIAL: NCT05321433
Title: The Association Between Tobacco Use and COVID-19 Infection and Adverse Outcomes in Three Nordic Countries: a Pooled Analysis
Brief Title: Tobacco Use and the Risk of COVID-19 and Adverse Outcomes
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government); Norwegian Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Maria Rosaria Galanti, Adjunct professor, Karolinska Institutet
Other Study IDs: 105544
Record Dates: First submitted 2022-04-08; First posted 2022-04-11 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Respiratory Tract Infections; Infections; Pneumonia, Viral; Pneumonia; Virus Diseases; SARS-CoV-2 Infection
Keywords: Tobacco; COVID-19; Snus; Epidemiology; Cohort Studies; Incidence
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections; Infections; Pneumonia, Viral; Pneumonia; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 11 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The Swedish Cohort: Swedish data comes from a historical cohort of 424,386 clients of public dental clinics aged 23 and older in the Stockholm region with inception between October 2015 and January 2020, with follow-up from February 2020 to December 2020. In Sweden, the public dental clinics (Folktandvården, FTV) provide routine preventive visits (oral check-ups) to all residents who choose to receive care in these clinics. At each health check-up smoking and snus use are ascertained as past use, current use, and amount of current use. The national personal numbers assigned to every resident in Sweden at birth or at immigration will be used to obtain information on diagnoses of COVID-19 and of other diseases through record-linkage with regional health care registers. Demographic information will be extracted through record-linkage with the register of the total population of the Stockholm region held by Statistics Sweden.
- The Finnish Cohort: The Finnish data will come from three pooled cross-sectional national health surveys in Finland (FinSote 2018-2020) of 44,199 participants aged 20 and older. The study samples included permanent residents in Finland from the FinSote surveys 2018, 2019, and 2020. The unique personal identifier assigned to all Finnish residents will be linked to the Communicable Diseases Registry to obtain information on diagnoses of COVID-19, to the Care Register for Health Care (HILMO) to obtain information on hospital admissions due to COVID-19, and to Statistics Finland Mortality Data to obtain information on deaths. Data on some sociodemographic characteristics will be also obtained from the Digital and Population Data Services Agency.
- The Norwegian Cohort: The Norwegian data will be based on the Norwegian Mother, Father and Child Cohort Study (MoBa) (Magnus et al., 2016), and the Norwegian Influenza Pregnancy Cohort (NorFlu) (Laake, 2018), with linkages to the Norwegian Surveillance System for Communicable Diseases (MSIS), the Norwegian Immunisation Registry (SYSVAK), and the Norwegian Population Registry. MoBa is a nation-wide population-based cohort consisting of 280 000 participants, where parents were recruited during pregnancy from 1999 to 2008, while NorFlu is a pregnancy cohort consisting of 9 000 participants recruited in Oslo and Bergen during the swine flu pandemic in 2009-2010. Demographic information is extracted from the registries via linkage to the existing cohort databases. For the purpose of this study, all subjects who died before the onset of the pandemic (February 2020) in the three countries will be excluded from the analysis.

SUMMARY:
This is an observational study of pooled population-based samples in three Nordic countries. Country-specific data has already been analysed in previous studies in Sweden, Finland, and Norway. The primary objective is to examine the association between tobacco use, the risk of SARS-CoV-2 infection, and adverse Outcomes using pooled population-based samples.

DETAILED DESCRIPTION:
The coronavirus disease (COVID-19) pandemic, caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), has caused more than 470 million confirmed cases of COVID-19, and more than 6 million deaths around the world by March 25, 2022 (WHO, 2022). Since the beginning of the COVID-19 pandemic, several factors have been attributed to increasing the risk of infection and adverse outcomes of the COVID-19 disease. Among these factors, the relationship between tobacco use and COVID-19 infection and adverse disease outcomes remained controversial as studies kept reporting mixed findings. Early studies reported what seemed to be a protective effect of tobacco use on COVID-19 infection (Haddad et al.; Jiménez-Ruiz et al., 2020), or hospitalizations due to COVID-19 (Farsalinos et al., 2020; Neira et al., 2021). A more recent ongoing living rapid review, this time including a larger selection of studies with different study designs, found that smokers are at reduced risk of SARS-COVID-19 infection compared to non-smokers (Relative risk 0.67, 95% Credible interval 0.60-0.75) (Simons et al., 2021). These findings opened the way for speculations and hypotheses on the potential mechanisms behind this protective role. However, results from most of these studies may be affected by selection bias as they reported findings from clinical samples or bias due to confounding as the structure of these published data permitted only univariate analysis.

Results from studies that suffer from selection bias or bias due to confounding should be handled with caution as they may undermine years of public health education against tobacco use, a major cause of morbidity and mortality worldwide. Moreover, the role of tobacco use in disease progression such as disease requiring hospitalization, ICU, and death remains unclear as most of the previous studies focused more on the association between tobacco use and the risk of infection, but not the adverse outcomes. These facts call for studies that ensure addressing any knowledge gap on the relation between tobacco and COVID-19 by taking into consideration 1) decreasing the risk for confounding and selection bias; 2) increasing precision through a higher sample size, 3) further investigating the association between tobacco use and adverse disease outcomes. In most Nordic countries, the profile of tobacco use in the underlying populations allows the analysis of several types of tobacco use e.g. cigarette smoking and smokeless tobacco (snus) use, enabling further insights into the potential role of nicotine in the association between tobacco use and COVID-19. The use of smokeless tobacco is highly prevalent (even exceeding the prevalence of smoking among men in Sweden and Norway), which will allow us to disentangle a potential role of nicotine in the association between tobacco use and COVID-19.

The investigators propose to examine the associations between tobacco use, COVID-19 infection, and adverse disease outcomes by using pooled population-based data from three Nordic countries, adjusting for potential confounders. The population-based nature of the samples minimizes selection bias Using a pooled analysis will accrue a large sample size and increase the potential for well-powered sub-groups analyses.

ELIGIBILITY:
Exclusion Criteria:

• All subjects who died before the onset of the pandemic (February 2020) in the three countries will be excluded from the analysis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational study of pooled population-based samples in three Nordic countries. Country-specific data has already been analysed in previous studies in Sweden (Galanti, 2021), Finland (Peña et al., 2021), and Norway (Magnus et al., 2016). We will use the national personal number assigned to every resident in these three countries at birth or at immigration to obtain information on diagnoses of COVID-19 and adverse outcomes among individuals in these cohorts through record-linkage with regional and national databases.
Sampling Method: Non-Probability Sample
Enrollment: 757585 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Any diagnosis of COVID-19 measured as follows: | February 2020 - December 2020
  Sweden: at least a positive polymerase chain reaction test (PCR) reported by the laboratories to Sweden's national electronic surveillance system for communicable diseases (SmiNet).
  Finland: cases with a positive SARS-CoV-2 reverse transcription PCR (RT-PCR), either informed by a laboratory or by a physician as a record of an International Classification of Diseases, Tenth Revision (ICD-10) code U07.1 (which requires a positive SARS-CoV-2 RT-PCR).
  Norway: a positive test for SARS-CoV-2 based on PCR obtained from The Norwegian Surveillance System for Communicable Diseases (MSIS) or the presence of antibodies for SARS-CoV-2.
  Out of these definitions a categorical variable will be created (No recorded COVID-19 diagnosis= 1, registered COVID-19 diagnosis= 2)
Hospital admission for COVID-19 measured as follows: | February 2020 - December 2020
  Any hospital admission with a diagnosis of COVID-19 (ICD-10 codes U071 and U072). The diagnosis could be registered either as a main or as a concomitant diagnosis.
  A. A categorical variable for hospital admission with any diagnosis of COVID-19 (either main or secondary diagnosis) will be created (No admissions= 1, any admission= 2).
  B. A categorical variable for hospital admission with COVID-19 as the main diagnosis only (No admissions= 1, any admission= 2).
Intensive unit care because of a diagnosis of COVID-19 measures as follows: | February 2020 - December 2020
  Admission to an intensive care unit (ICU) because of a diagnosis of COVID-19 (ICD-10 codes as above). A categorical variable for intensive unit care because of a diagnosis of COVID-19 (No/Yes) will be created (No ICU care= 1, any ICU care= 2).
Death for COVID-19 measured as follows: | February 2020 - December 2020
  Death due to COVID-19 will be established using the Swedish, Finnish, and Norwegian Cause of Death Registries. All deaths occurring during the follow-up period with COVID-19 registered as the main cause will be included.

SECONDARY OUTCOMES:
Length of hospital stay for COVID-19 | February 2020 - December 2020
  As a secondary analysis, we will use a negative binomial count model (Hilbe, 2011, 2014) to assess inpatient length of stay measured as the cumulative number of days of hospitalization, as an indicator of disease severity among tobacco users compared to non-tobacco users.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosaria Galanti, Principal Investigator — Department of Global Public Health, Karolinska Institute
Locations (1):
- Karolinska Institutet, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen PK, Abildstrom SZ, Rosthoj S. Competing risks as a multi-state model. Stat Methods Med Res. 2002 Apr;11(2):203-15. doi: 10.1191/0962280202sm281ra. PMID 12040697
- [Background] Austin PC, Lee DS, Fine JP. Introduction to the Analysis of Survival Data in the Presence of Competing Risks. Circulation. 2016 Feb 9;133(6):601-9. doi: 10.1161/CIRCULATIONAHA.115.017719. PMID 26858290
- [Background] Berry SD, Ngo L, Samelson EJ, Kiel DP. Competing risk of death: an important consideration in studies of older adults. J Am Geriatr Soc. 2010 Apr;58(4):783-7. doi: 10.1111/j.1532-5415.2010.02767.x. Epub 2010 Mar 22. PMID 20345862
- [Background] Farsalinos, K., Barbouni, A., & Niaura, R. (2020). Smoking, vaping and hospitalization for COVID-19. Qeios.
- [Background] Fine, J. P., & Gray, R. J. (1999). A proportional hazards model for the subdistribution of a competing risk. Journal of the American Statistical Association, 94(446), 496-509.
- [Background] Galanti, M. R. (2021). Tobacco Use and the Risk of COVID-19. ClinicalTrials.gov: NCT04896918. 2021. [Available from: https://clinicaltrials.gov/ct2/show/NCT04896918].
- [Background] Goldstein, H. (1995). Multilevel Statistical Models, Chapter 2. Edward Arnold. In: London, Wiley, New York.
- [Background] Haddad C, Bou Malhab S, Sacre H, Salameh P. Smoking and COVID-19: A Scoping Review. Tob Use Insights. 2021 Feb 15;14:1179173X21994612. doi: 10.1177/1179173X21994612. eCollection 2021. PMID 33642886
- [Background] Hilbe, J. M. (2011). Negative binomial regression. Cambridge University Press.
- [Background] Hilbe, J. M. (2014). Modeling count data. Cambridge University Press.
- [Background] Ioannidis JPA. Over- and under-estimation of COVID-19 deaths. Eur J Epidemiol. 2021 Jun;36(6):581-588. doi: 10.1007/s10654-021-00787-9. Epub 2021 Jul 28. PMID 34322831
- [Background] Jimenez-Ruiz CA, Lopez-Padilla D, Alonso-Arroyo A, Aleixandre-Benavent R, Solano-Reina S, de Granda-Orive JI. [COVID-19 and Smoking: A Systematic Review and Meta-Analysis of the Evidence]. Arch Bronconeumol. 2021 Jan;57:21-34. doi: 10.1016/j.arbres.2020.06.024. Epub 2020 Jul 25. Spanish. PMID 34629638
- [Background] Kim HT. Cumulative incidence in competing risks data and competing risks regression analysis. Clin Cancer Res. 2007 Jan 15;13(2 Pt 1):559-65. doi: 10.1158/1078-0432.CCR-06-1210. PMID 17255278
- [Background] Laake I, Tunheim G, Robertson AH, Hungnes O, Waalen K, Haberg SE, Mjaaland S, Trogstad L. Risk of pregnancy complications and adverse birth outcomes after maternal A(H1N1)pdm09 influenza: a Norwegian population-based cohort study. BMC Infect Dis. 2018 Oct 22;18(1):525. doi: 10.1186/s12879-018-3435-8. PMID 30348103
- [Background] Magnus P, Birke C, Vejrup K, Haugan A, Alsaker E, Daltveit AK, Handal M, Haugen M, Hoiseth G, Knudsen GP, Paltiel L, Schreuder P, Tambs K, Vold L, Stoltenberg C. Cohort Profile Update: The Norwegian Mother and Child Cohort Study (MoBa). Int J Epidemiol. 2016 Apr;45(2):382-8. doi: 10.1093/ije/dyw029. Epub 2016 Apr 10. PMID 27063603
- [Background] Puebla Neira D, Watts A, Seashore J, Polychronopoulou E, Kuo YF, Sharma G. Smoking and risk of COVID-19 hospitalization. Respir Med. 2021 Jun;182:106414. doi: 10.1016/j.rmed.2021.106414. Epub 2021 Apr 17. PMID 33915414
- [Background] Peña, S., Ilmarinen, K., Kestilä, L., & Karvonen, S. (2021). Tobacco Use and COVID-19 Incidence in the Finnish General Population (Tobrisk-CoV). ClinicalTrials.gov: NCT04915781. 2021. [Available from: https://clinicaltrials.gov/ct2/show/NCT04915781]. https://clinicaltrials.gov/ct2/show/NCT04915781
- [Background] Simons D, Shahab L, Brown J, Perski O. The association of smoking status with SARS-CoV-2 infection, hospitalization and mortality from COVID-19: a living rapid evidence review with Bayesian meta-analyses (version 7). Addiction. 2021 Jun;116(6):1319-1368. doi: 10.1111/add.15276. Epub 2020 Nov 17. PMID 33007104
- [Background] Southern DA, Faris PD, Brant R, Galbraith PD, Norris CM, Knudtson ML, Ghali WA; APPROACH Investigators. Kaplan-Meier methods yielded misleading results in competing risk scenarios. J Clin Epidemiol. 2006 Oct;59(10):1110-4. doi: 10.1016/j.jclinepi.2006.07.002. PMID 16980152
- [Background] WHO. (2022). Coronavirus (COVID-19) Dashboard. https://covid19.who.int/]
- [Background] Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702-6. doi: 10.1093/aje/kwh090. PMID 15033648
- See also: Tobacco Use and the Risk of COVID-19. ClinicalTrials.gov: NCT04896918. — https://clinicaltrials.gov/ct2/show/NCT04896918
- See also: Tobacco Use and COVID-19 Incidence in the Finnish General Population (Tobrisk-CoV). ClinicalTrials.gov: NCT04915781. — https://clinicaltrials.gov/ct2/show/NCT04915781

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT05321433/Prot_SAP_000.pdf